CLINICAL TRIAL: NCT03418857
Title: The Role of Probiotics in Attenuating Inflammation and Improving Gut Health in Obese Adults
Brief Title: Probiotics and Gut Health
Acronym: PRO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Connie J Rogers, Associate Professor of Nutritional Sciences, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY0006843
Record Dates: First submitted 2017-12-13; First posted 2018-02-01 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Metabolic Syndrome
Keywords: probiotics; Human; obesity; non-pharmacologic therapy; gut health; microbiome; inflammation
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants will consume one yogurt smoothie daily for the duration of the intervention that contains 3.16 × 109 colony forming units (CFU) bifidobacterium animalis subsp. lactis BB-12. Participants will be asked to refrain from consumption of other yogurt or probiotic-containing foods.
  Interventions: Drug: Yogurt smoothie with BB-12
- Control (Placebo Comparator): Participants will consume one yogurt smoothie daily for the duration of the intervention that contains no BB-12. Participants will be asked to refrain from consumption of other yogurt or probiotic-containing foods.
  Interventions: Drug: Yogurt smoothie

INTERVENTIONS:
Drug: Yogurt smoothie with BB-12 — During the one month intervention period, the participants will consume one yogurt smoothie with BB-12 daily.
  Arms: Experimental
Drug: Yogurt smoothie — During the one month control period, the participants will consume one yogurt smoothie daily.
  Arms: Control

SUMMARY:
This study evaluates the effects of probiotic consumption on inflammatory outcomes and measures of gut health. Participants will be given yogurt with probiotics for one period and yogurt without probiotics for another, with a break in between. These periods will occur in random order.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ to 25 and less than 35 kg/m^2
* Increased waist circumference (men: ≥ 94 cm, women: ≥ 80 cm)
* At least one of the metabolic syndrome criteria-
* serum triglycerides: ≥ 150 mg/dL
* HDL cholesterol: ≤ 40 mg/dL in men, ≤ 50 mg/dL in women
* blood pressure: ≥ 130 mmHg systolic or ≥ 85 mmHg diastolic
* fasting plasma glucose ≥ 100 mg/dL

Exclusion Criteria:

* allergy to dairy
* smoking and/or use of tobacco products
* systolic blood pressure ≥ 160 mmHg
* diastolic blood pressure > 100 mmHg
* fasting glucose ≥ 126 mg/dL
* history of myocardial infarction, cardiovascular disease (CVD), stroke, diabetes mellitus, liver disease, kidney disease, thyroid disease (unless controlled on medication)
* use of cholesterol or lipid lowering medications
* use of anti-hypertensive or glucose lowering supplements (psyllium, fish oil capsules, soy lecithin, niacin, fiber, flax, phytoestrogens, and stanol/sterol supplemented foods)
* refusal to discontinue nutritional supplements, herbs, vitamins, or other probiotics
* clinical diagnosis of inflammatory bowel disease (IBD) e.g. Chron's disease or ulcerative colitis
* Use of antibiotics within the last 2 months
* excessive alcohol consumption (≥ 14 standard drinks per week)
* regular use of anti-inflammatory medications (e.g. aspirin, ibuprofen)

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-29 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in inflammatory markers | At baseline before intervention period 1, at endpoint of intervention period 1 (week 4), at baseline before intervention period 2 (week 8), at endpoint after intervention period 2 (week 12)
  Change in inflammatory markers in the serum and secreted cytokines from lipopolysaccharide (LPS)-stimulated peripheral blood mononuclear cells compared to baseline. In the serum the markers to be investigated are high sensitivity c-reactive protein (hs-CRP), tumor necrosis factor alpha (TNF-a), interleukin 1 beta (IL-1B), IL-6, IL-8, IL-10, IL-12p70, monocyte chemotactic protein 1 (MCP-1), macrophage inflammatory protein alpha (MIP-1a), sCD14, and LPS binding protein (LPB). From LPS-stimulated peripheral blood mononuclear cells the cytokines to be investigated are TNF-a, IL-1B, IL-6, IL-8, IL-10, IL-12p70, MCP-1, and MIP-1a. Changes in these inflammatory markers will assist in understanding how the consumption of yogurt containing BB-12 affects the inflammatory status of obese individuals.

SECONDARY OUTCOMES:
Change in number and activation of leukocytes | At baseline before intervention period 1, at endpoint of intervention period 1 (week 4), at baseline before intervention period 2 (week 8), at endpoint after intervention period 2 (week 12)
  Change in quantity and activation of T cells, B cells, dendritic cells, natural killer cells, and monocytes measured by flow cytometry before and after each period. Changes in the number and activation of leukocytes will assist in understanding the impacts of the consumption of yogurt containing BB-12 on leukocytes in obese individuals.
Change in gut permeability | At baseline before intervention period 1, at endpoint of intervention period 1 (week 4), at baseline before intervention period 2 (week 8), at endpoint after intervention period 2 (week 12)
  Change in gut permeability, assessed using a lactulose/mannitol gut permeability assay, from baseline. Changes in gut permeability will assist in understanding the impacts of the consumption of yogurt containing BB-12 on gut health and permeability in obese individuals.
Change in gut microbiota populations | At baseline before intervention period 1, at endpoint of intervention period 1 (week 4), at baseline before intervention period 2 (week 8), at endpoint after intervention period 2 (week 12)
  Change in gut microbiota populations, assessed with 16s ribosomal ribonucleic acid (rRNA), compared to baseline. Changes in microbial populations will assist in understanding the impacts of the consumption of yogurt containing BB-12 on commensal gut microbiota in obese individuals.
Change in metabolism of gut microbiota populations | At baseline before intervention period 1, at endpoint of intervention period 1 (week 4), at baseline before intervention period 2 (week 8), at endpoint after intervention period 2 (week 12)
  Change in the metabolism of gut microbiota populations, measured via transcriptomics, compared to baseline. Changes in the transcriptome of the commensal microbiota will assist in understanding the impacts of the consumption of yogurt containing BB-12 on the metabolism of commensal gut microbiota in obese individuals.

OTHER OUTCOMES:
Change in trimethylamine N-oxide (TMAO) in serum | At baseline before intervention period 1, at endpoint of intervention period 1 (week 4), at baseline before intervention period 2 (week 8), at endpoint after intervention period 2 (week 12)
  Change in TMAO in serum measured using liquid chromatography with tandem mass spectrometry (LC-MS) compared to baseline. Changes in TMAO, which is associated with gut microbiota, will assist in understanding the mechanism that connects changes in the commensal microbiota in the gut to inflammatory outcomes in obese individuals.
Change in serum metabolomic profile | At baseline before intervention period 1, at endpoint of intervention period 1 (week 4), at baseline before intervention period 2 (week 8), at endpoint after intervention period 2 (week 12)
  Change in serum metabolomic profile, assessed in hydrophilic and hydrophobic fractions, compared to baseline. Changes in the metabolomic profile will assist in understanding the underlying mechanisms that connect consumption of yogurt containing BB-12 to changes in inflammatory status in obese individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

REFERENCES:
- [Background] Meng H, Ba Z, Lee Y, Peng J, Lin J, Fleming JA, Furumoto EJ, Roberts RF, Kris-Etherton PM, Rogers CJ. Consumption of Bifidobacterium animalis subsp. lactis BB-12 in yogurt reduced expression of TLR-2 on peripheral blood-derived monocytes and pro-inflammatory cytokine secretion in young adults. Eur J Nutr. 2017 Mar;56(2):649-661. doi: 10.1007/s00394-015-1109-5. Epub 2015 Nov 30. PMID 26621631
- [Background] Aggarwal BB. Targeting inflammation-induced obesity and metabolic diseases by curcumin and other nutraceuticals. Annu Rev Nutr. 2010 Aug 21;30:173-99. doi: 10.1146/annurev.nutr.012809.104755. PMID 20420526
- [Background] Leber B, Tripolt NJ, Blattl D, Eder M, Wascher TC, Pieber TR, Stauber R, Sourij H, Oettl K, Stadlbauer V. The influence of probiotic supplementation on gut permeability in patients with metabolic syndrome: an open label, randomized pilot study. Eur J Clin Nutr. 2012 Oct;66(10):1110-5. doi: 10.1038/ejcn.2012.103. Epub 2012 Aug 8. PMID 22872030
- [Background] Cani PD, Bibiloni R, Knauf C, Waget A, Neyrinck AM, Delzenne NM, Burcelin R. Changes in gut microbiota control metabolic endotoxemia-induced inflammation in high-fat diet-induced obesity and diabetes in mice. Diabetes. 2008 Jun;57(6):1470-81. doi: 10.2337/db07-1403. Epub 2008 Feb 27. PMID 18305141
- [Background] Sugahara H, Odamaki T, Fukuda S, Kato T, Xiao JZ, Abe F, Kikuchi J, Ohno H. Probiotic Bifidobacterium longum alters gut luminal metabolism through modification of the gut microbial community. Sci Rep. 2015 Aug 28;5:13548. doi: 10.1038/srep13548. PMID 26315217
- [Background] Rizzardini G, Eskesen D, Calder PC, Capetti A, Jespersen L, Clerici M. Evaluation of the immune benefits of two probiotic strains Bifidobacterium animalis ssp. lactis, BB-12(R) and Lactobacillus paracasei ssp. paracasei, L. casei 431(R) in an influenza vaccination model: a randomised, double-blind, placebo-controlled study. Br J Nutr. 2012 Mar;107(6):876-84. doi: 10.1017/S000711451100420X. Epub 2011 Sep 7. PMID 21899798